CLINICAL TRIAL: NCT07205289
Title: A Phase 1B Open-label Study to Collect Serum Following Vaccination With Killed Whole-cell Pneumococcal Vaccine (Gamma-PN) in Adults for Use in Assay Validation
Brief Title: Serum Collection Study for Assay Development
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GPN Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GPNV-008
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Disease, Invasive; Pneumococcal Disease
Keywords: Vaccination pneumococcal
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamma -PN (Experimental): Intramuscular administration 500 mcg
  Interventions: Biological: Gamma-PN

INTERVENTIONS:
Biological: Gamma-PN — Killed whole-cell pneumococcal vaccine

SUMMARY:
The study will collect serum from 12 participants vaccinated with Gamma-PN to assist with assay development and validation

DETAILED DESCRIPTION:
The study will collect serum from 12 participants vaccinated with Gamma-PN to assist with assay development and validation

Participants will receive a dose of Gamma-PN and serum will be collected pre dose and Day 28

ELIGIBILITY:
Inclusion Criteria:

* good general health

Exclusion Criteria:

* no previous pneumococcal vaccine

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
OPA | 6 months
  Opsonophagocytic assay

CONTACTS AND LOCATIONS:
Overall Officials: Eve Kennedy, PhD, Study Director — GPN Vaccines Ltd
Locations (1):
- University of Adelaide Clinical Research Facility, Adelaide, South Australia, Australia